CLINICAL TRIAL: NCT00001997
Title: Safety and Efficacy of Polyethylene Glycolated IL-2 (PEG IL-2) Plus Zidovudine or Dideoxyinosine in HIV Positive, Asymptomatic and Symptomatic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 072B; CS-PG91-07
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1991-07

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Polyethylene Glycols; Interleukin-2; Didanosine; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Interleukin-2, Polyethylene Glycolated
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To investigate the safety of polyethylene glycolated interleukin-2 (PEG IL-2) given subcutaneously in conjunction with antiviral treatment and to explore the effects of treatment on surrogate markers of efficacy and incidence of opportunistic infection and other clinical markers of HIV disease.

DETAILED DESCRIPTION:
Four escalating doses of PEG IL-2 are studied. Patients are stratified by CD4 level. CD4 levels in Group A are 200 to 500 cells/mm3; in Group B - 1 to less than 200 cells/mm3. Further stratification is by p24 positive or negative, antiviral therapy for more or less than a year, and zidovudine (AZT) versus didanosine (ddI). The duration of PEG IL-2 treatment is a maximum of 28 weeks. This is an outpatient study; patients will be observed for four hours after the first dose of PEG IL-2 and for one hour after subsequent doses.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity by commercially available ELISA.
* Meet Disease Status criteria.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Concurrent neoplasms other than basal cell carcinoma of the skin, in-situ carcinoma of the cervix or limited cutaneous Kaposi's sarcoma.
* Recently treated HIV-related lymphoma.
* Major organ allograft.
* Presence of space occupying central nervous system (CNS) lesions or other conditions which would be anticipated to cause cerebral edema.
* Renal compromise or use of drug therapy anticipated to lead to renal compromise.
* Active opportunistic infection requiring hospitalization or exclude medication.
* Requiring continual acyclovir for suppression of herpes infection.

Concurrent Medication:

Excluded:

* Acyclovir.
* Drug therapy anticipated to lead to renal compromise.

Patients with the following are excluded:

* Intolerance to zidovudine (AZT) at 300 mg/day divided q8h or didanosine (ddI) at 7 mg/kg/day given twice a day.
* History of HIV-related lymphoma.
* History of asthma requiring frequent therapy, chronic pulmonary disease, hypertension requiring therapy, or congestive heart failure.
* Any of the symptoms or conditions listed in Exclusion - Co-Existing Conditions.

Prior Medication:

Excluded:

- Any prior therapy with interleukin-2 (IL-2) or PEG IL-2.

Excluded 30 days prior to study entry:

- Treatment with other anti-HIV medication or known immunomodulators or other chemotherapy or radiation therapy.

Active substance abuse so patients would be anticipated to be poorly compliant with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Dr David R Senechek, San Francisco, California, United States